CLINICAL TRIAL: NCT04140903
Title: Partial Oral Antibiotic Treatment for Bacterial Brain Abscess: an Open-label Randomised Non-inferiority Trial
Brief Title: Partial Oral Antibiotic Treatment for Bacterial Brain Abscess
Acronym: ORAL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henrik Nielsen (Other)
Responsible Party: Sponsor-Investigator, Henrik Nielsen, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2019-07-04; First posted 2019-10-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Brain Abscess; Cerebral Abscess
Keywords: Oral antibiotics
MeSH Terms: conditions — Brain Abscess

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, international, multi-centre, randomised, parallel groups, non-inferiority trial
Who Masked: Outcomes Assessor
Masking Description: An independent blinded endpoint committee will assess the primary outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral antibiotics (Experimental): Patients will be randomised to oral antibiotics after two weeks of appropriate antibiotic therapy for bacterial brain abscess since definitive aspiration/excision of brain abscess or, in case of no planned diagnostic neurosurgical procedure, since initiation of guideline recommended antibiotics for bacterial brain abscess
  Interventions: Drug: Early transition to oral antibiotics
- Standard treatment (Active Comparator): Patients will be randomised to continuation of standard intravenous antibiotics after two weeks of appropriate antibiotic therapy for bacterial brain abscess since definitive aspiration/excision of brain abscess or, in case of no planned diagnostic neurosurgical procedure, since initiation of guideline recommended antibiotics for bacterial brain abscess
  Interventions: Drug: Standard treatment of intravenous antibiotics

INTERVENTIONS:
Drug: Early transition to oral antibiotics — Patients will be treated with an oral antibiotic regimen (e.g. amoxicillin + metronidazole) based upon pharmacokinetic and pharmacodynamic properties of the drugs, pathogen susceptibility, and any existing drug allergies or interactions
  Arms: Oral antibiotics
Drug: Standard treatment of intravenous antibiotics — Patients will continue standard intravenous antibiotic therapy for brain abscess (e.g. 3rd generation cephalosporin + metronidazole) according to international guidelines and pathogen susceptibility patterns.
  Arms: Standard treatment

SUMMARY:
The investigators aim to determine if oral antibiotics are clinically acceptable as treatment of brain abscess. Following 2 weeks of standard intravenous antibiotic therapy, half of patients will continue with this treatment for another 4 weeks or longer while the other half will be assigned to oral antibiotics for the remaining duration of treatment.

DETAILED DESCRIPTION:
Treatment of brain abscess remains a considerable challenge due to the precarious location of the infection and the impenetrability of the blood-brain-barrier for most drugs. Thus, cure usually requires a combination of neurosurgical evacuation of abscess material and 6-8 weeks of high-dose intravenous (IV) antibiotic therapy to ensure eradication of bacteria within the abscess cavity. Disadvantages include risks of nosocomial infections and line-associated complications (e.g. bleeding, venous thrombosis, or need for replacement due to malfunction) in addition to the considerable costs of such long-term admission. However, improved insights into the pharmacokinetic properties and favourable bioavailability of some oral antibiotics may allow such treatment at an early stage. To date, there are no randomised controlled trials to guide treatment of bacterial brain abscess.

The investigators wish to determine whether a treatment strategy of transition to oral antibiotics after two weeks of treatment is non-inferior to continued IV antibiotics in clinically stable brain abscess patients assessed by the proportion with a favourable outcome at six months since randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical presentation (e.g. headache, neurological deficit or fever) and cranial imaging (CT or MRI) consistent with brain abscess AND
2. The physician responsible for the patient decides to treat the patient for bacterial brain abscess AND
3. Ability to take and absorb oral medications (including by nasogastric tube) AND
4. To have received relevant antibiotic therapy for bacterial brain abscess for 14 consecutive days before randomisation AND
5. Expected to be treated with antibiotic therapy for at least another 14 days after time of randomisation AND
6. No progression in symptom intensity or occurrence of new-onset neurological symptoms (excluding seizures) within five days before time of randomisation.

Exclusion Criteria (patients fulfilling either criteria):

1. Expected substantially reduced compliance with treatment (e.g. IV drug abuse)
2. Pregnancy (proven by positive urine or plasma human chorionic gonadotropin test in fertile women <50 years of age)
3. Concomitant (empirical) brain abscess treatment for tuberculosis, nocardiosis, Pseudomonas spp., fungi, toxoplasmosis or other CNS parasites
4. Device related brain abscesses (e.g. deep brain stimulators, ventriculo-peritoneal shunts)
5. Severe immuno-compromise defined as ongoing need for biological- or chemotherapy, prednisolone >20 mg/day for 14 days or longer, uncontrolled HIV/AIDS, haematological malignancies, and organ transplant recipients
6. Concomitant or unrelated infections necessitating IV antibiotics beyond seven days of duration after time of randomisation
7. Previous enrolment into this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | Six months after randomisation
  A composite of number of participants with all-cause mortality, risk of intraventricular rupture of brain abscess (IVROBA), unplanned neurosurgery, relapse, or recurrence

SECONDARY OUTCOMES:
Treatment failure | At last day of antibiotic treatment for brain abscess, and 3- and 12-months after randomisation
  A composite of number of participants with all-cause mortality, risk of intraventricular rupture of brain abscess (IVROBA), unplanned neurosurgery, relapse, or recurrence
Unfavourable outcome | At last day of antibiotic treatment for brain abscess, and 3-, 6-, and 12-months after randomisation
  Number of participants with Extended Glasgow Outcome Scale score <7, overall and stratified by study centre, oral cavity bacteria (yes/no) and largest brain abscess diameter (+/- 3 cm)
All-cause mortality | At last day of antibiotic treatment for brain abscess, and 3-, 6-, and 12-months after randomisation
  Number of participants with fatal outcome, overall and stratified by study centre, oral cavity bacteria (yes/no) and largest brain abscess diameter (+/- 3 cm)
Unplanned neurosurgery | At 6 months since randomisation
  Number of participants with unplanned (re-)aspiration or excision, overall and stratified by study centre, oral cavity bacteria (yes/no) and largest brain abscess diameter (+/- 3 cm)
IVROBA | At 6 months since randomisation
  Number of participants with intraventricular rupture of brain abscess, overall and stratified by study centre, oral cavity bacteria (yes/no) and largest brain abscess diameter (+/- 3 cm)
Relapse | At 6 months since randomisation
  Number of participants with increase in brain abscess volume by 20% since randomisation, clinical deterioration attributable to brain abscess or lack of cure of at least 4 weeks or longer of assigned study treatment, overall and stratified by study centre, oral cavity bacteria (yes/no) and largest brain abscess diameter (+/- 3 cm)
Recurrence | At 6 months since randomisation
  New brain abscess formation after end of treatment, overall and stratified by study centre, oral cavity bacteria (yes/no) and largest brain abscess diameter (+/- 3 cm)
Unfavourable outcome - sliding dichotomy | At last day of antibiotic treatment for brain abscess, and 3-, 6-, and 12-months after randomisation
  Sliding dichotomy of extended Glasgow Outcome Scale scores according to Charlson comorbidity index score (range: 0=no comorbidity and more likely to have a favourable outcome to 40=high degree of comorbidity with a poor prognosis of a favourable outcome) at time of randomisation (0 vs. 1-2 vs. >2).
Central line associated complications | 6 months since randomisation
  Number of participants with bleeding, infection, venous thrombosis or need for replacement of central line due to mechanical malfunction
Clostridial diarrhea | From randomisation up until last day antibiotic treatment for brain abscess
  Number of participants who develop Clostridioides difficile associated gastro-enteritis during antibiotic treatment for brain abscess
Duration of admission | From randomisation until hospital discharge to home or rehabilitation unit or death, whichever comes first, assessed up to 6 months
  Days spent as admitted patient in hospital up to 6 months since randomisation (does not include outpatient hospital care)
Duration of treatment | From randomisation until last day of antibiotic treatment for brain abscess up to 6 months since randomisation
  Number of days treated with antibiotics for brain abscess up to 6 months since randomisation
Adherence to treatment | From randomisation until last day of antibiotic treatment for brain abscess, assessed up to 6 months since randomisation
  Adherence to allocated treatment. For oral treatment this will be measured using Morisky 8-item Medication Adherence scale scores (range 0=high adherence to 8=low adherence) up to 6 months since randomisation
Oedema on cranial imaging | 3 months since randomisation
  Number of participants with residual perilesional oedema on cranial imaging up to 3 months since randomisation
SAE | From randomisation until last day of antibiotic treatment for brain abscess
  Number of participants with severe adverse events
SF36 | At time of randomisation, last day of antibiotic treatment for brain abscess, and 3-, 6-, and 12-months since randomisation
  Short Form 36 is a 36 item survey of patient-reported health-related quality of life (range 0=maximum disability to 100=no disability)
EQ-5D-5L | At time of randomisation, last day of antibiotic treatment for brain abscess, and 3-, 6-, and 12-months since randomisation
  EuroqQol - 5 dimensions - 5 level scores are derived from a standardized instrument for measuring generic health status including mobility, self-care, usual acitivities, pain/discomfort, and anxiety/depression (range 5=good health status to 25=poor health status)
EQ-VAS | At time of randomisation, last day of antibiotic treatment for brain abscess, and 3-, 6-, and 12-months since randomisation
  EuroqQol Visual Analogue Scale (range 0=poor health status to 100=excellent health status)
Cognitive impairment | At time of randomisation, last day of antibiotic treatment for brain abscess, and 3-, 6-, and 12-months since randomisation
  Montreal Cognitive Assessment (MoCA) scores (range 0=poor cognitive performance to 30=normal cognitive performance)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bodilsen, MD, Principal Investigator — Aalborg University Hospital
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
Beginning six months and ending three years after publication, an anonymized dataset can be shared with qualified researchers who provide a methodologically sound proposal for a post-hoc study assessed by the members of the steering committee. The anonymized dataset will include baseline demographics of patients, laboratory results, treatments and primary outcome at six months since randomisation. In addition, the study protocol, statistical analysis plan, informed consent form, clinical study report and analytic code can also be shared. Proposals should be directed to the trial manager. To gain access, data requestors will need to sign a data access agreement. Data will be deposited at Mendeley Data (https://data.mendeley.com/).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months until 3 years after publication
Access Criteria: Qualified researchers who provide a methodologically sound proposal for a post-hoc study assessed by the members of the steering committee may gain access to data after proper governmental approvals have been obtained.
URL: https://data.mendeley.com

REFERENCES:
- [Derived] Bodilsen J, Brouwer MC, van de Beek D, Tattevin P, Tong S, Naucler P, Nielsen H. Partial oral antibiotic treatment for bacterial brain abscess: an open-label randomized non-inferiority trial (ORAL). Trials. 2021 Nov 12;22(1):796. doi: 10.1186/s13063-021-05783-8. PMID 34772441